CLINICAL TRIAL: NCT00833677
Title: Community Based Participatory Research With Immigrant Chinese With Type 2 Diabetes: Adapting and Testing Coping Skills Training.
Brief Title: Community Based Participatory Research With Immigrant Chinese With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of San Francisco (Other); Donaldina Cameron House (Unknown); North East Medical Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H2269-32042-02; 1R01NR010693-01 (NIH)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Coping skills; Chinese; Immigrant; Type 2 Diabetes Mellitus; Family research
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Chinese Coping Skills Training — Six-week group behavioral intervention: Chinese Coping Skills Training

SUMMARY:
The proposed project is part of a program of research to improve management of type 2 diabetes (T2DM) through a community-academic partnership that addresses cultural factors in disease management. Specific aims are to: 1. Strengthen a community-academic partnership with the immigrant Chinese community in San Francisco to improve diabetes management; 2. Adapt and test a behavioral diabetes intervention, Coping Skills Training, to addresses family and cultural issues in immigrant Chinese patients with T2DM; and 3. Disseminate the adapted Coping Skills Training Program findings via the community-academic partnership to the immigrant Chinese American community through service programs, ethnic media, and professional/scientific publications. A mixed-methods CBPR approach will be used to interpretively adapt a behavioral intervention to be culturally appropriate, and test its efficacy using a repeated measures design. Two historically significant social service and health agencies serving immigrant Chinese in San Francisco are collaborating with this nurse-led interdisciplinary research team.

DETAILED DESCRIPTION:
The goal of the culturally adapted Chinese Coping Skills Training (CCST) is to increase immigrant Chinese patients' skills and mastery in diabetes management by identifying and diminishing non-constructive coping responses to difficult social situations, while expanding the repertoire of positive coping responses and disease management behaviors. The CCST comprises a series of six small-group sessions focused on the topics of social problem solving, communication skills, cognitive behavior modification and conflict resolution. It also includes a review of basic diabetes management information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus,
* Treated with insulin, oral medications and/or diet and exercise,
* Self-identify as Chinese American or Chinese,
* Identify a family member (spouse, child, sibling or other person identified as family) with whom participant lives or has at least weekly contact, who is involved in care of diabetes.
* First-generation immigrant ie. foreign-born, first generation to arrive in the U.S. from any source country

Exclusion Criteria:

* Diagnosed with type 1 diabetes mellitus
* Cannot read or write Chinese

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Diabetes Self Efficacy | 16 weeks post treatment-as compared with the delayed-treatment phase.

SECONDARY OUTCOMES:
Diabetes Specific Conflict | 16 weeks post treatment as compared with the delayed treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chesla, DNS, Principal Investigator — University of California, San Francisco
Locations (1):
- School of Nursing, University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Chesla CA, Chun KM. Accommodating type 2 diabetes in the Chinese American family. Qual Health Res. 2005 Feb;15(2):240-55. doi: 10.1177/1049732304272050. PMID 15611206
- [Background] Fisher L, Chesla CA, Chun KM, Skaff MM, Mullan JT, Kanter RA, Gardiner PS. Patient-appraised couple emotion management and disease management among Chinese American patients with type 2 diabetes. J Fam Psychol. 2004 Jun;18(2):302-10. doi: 10.1037/0893-3200.18.2.302. PMID 15222837
- [Background] Chesla CA, Chun KM, Kwan CM. Cultural and family challenges to managing type 2 diabetes in immigrant Chinese Americans. Diabetes Care. 2009 Oct;32(10):1812-6. doi: 10.2337/dc09-0278. Epub 2009 Jul 23. PMID 19628812
- [Background] Chun KM, Chesla CA, Kwan CM. "So We Adapt Step by Step": Acculturation experiences affecting diabetes management and perceived health for Chinese American immigrants. Soc Sci Med. 2011 Jan;72(2):256-64. doi: 10.1016/j.socscimed.2010.11.010. Epub 2010 Nov 24. PMID 21147509